CLINICAL TRIAL: NCT00988429
Title: Efficacy and Safety of Eslicarbazepine Acetate (BIA 2-093) as Adjunctive Therapy for Refractory Partial Seizures in a Double-blind, Randomised, Placebo-controlled, Parallel-group, Multicentre Trial
Brief Title: Efficacy and Safety of Eslicarbazepine Acetate (BIA 2-093) as Adjunctive Therapy for Refractory Partial Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIA-2093-304; 2008-002455-25 (EudraCT Number)
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Results first posted 2014-04-15 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2018-10

CONDITIONS: Partial Epilepsy
Keywords: Refractory; partial; epilepsy; efficacy; eslicarbazepine; safety
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 800 mg QD Eslicarbazepine acetate (Active Comparator): tablets
  Interventions: Drug: 800 mg QD Eslicarbazepine acetate
- 1200 mg QD Eslicarbazepine acetate (Active Comparator): tablets
  Interventions: Drug: 1200 mg QD Eslicarbazepine acetate
- Placebo (Placebo Comparator): tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 800 mg QD Eslicarbazepine acetate — Oral, 800 mg QD, 2-week titration period and 12-week maintenance period
  Other Names: BIA 2-093
  Arms: 800 mg QD Eslicarbazepine acetate
Drug: 1200 mg QD Eslicarbazepine acetate — Oral, 1200 mg QD, 2-week titration followed by 12-week maintenance period
  Other Names: BIA 2-093
  Arms: 1200 mg QD Eslicarbazepine acetate
Drug: Placebo — Placebo tablet given QD
  Other Names: Sugar pills
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Eslicarbazepine acetate (BIA 2-093) is an effective adjunct therapy in the treatment of refractory partial seizures

DETAILED DESCRIPTION:
The study was designed to include 3 parts; only the first part is described in this report. Part I of the study was an international, randomized, placebo-controlled, double-blind, parallel group, multicenter clinical study conducted in 19 countries at 173 sites in 653 subjects with refractory simple partial or complex partial seizures, with or without secondary generalization. After screening procedures and confirming eligibility, subjects entered Part I of the study, which consisted of 3 periods.

The first period was an 8 week observation baseline period (Week -8 to Week -1) during which subjects were instructed on how to complete the seizure diary. At the end of the 8 week observational baseline period, eligible subjects were randomized in a 1:1:1 allocation ratio to 1 of 3 treatment groups (with a blinded treatment assignment):

* Placebo
* ESL 800 mg QD
* ESL 1200 mg QD Subjects then entered the second period of Part 1, the 2 week, double blind, up titration period (Week 1 to Week 2). During this period, subjects in the ESL 800 mg group received ESL 400 mg QD, subjects in the ESL 1200 mg group received ESL 800 mg QD, and subjects in the placebo group received placebo QD.

Subjects then entered the third period of Part I, the 12 week, double-blind, maintenance period (Week 3 to Week 14) where subjects in the ESL 800 mg group received ESL 800 mg QD, subjects in the ESL 1200 mg group received ESL 1200 mg QD, and subjects in the placebo group received placebo QD.

At the completion of the maintenance period, subjects who did not enter Part II were to be tapered off study drug while maintaining the blind according to the following down titration procedure: subjects on 800 mg were down titrated to 400 mg for a duration of 2 weeks, and subjects on 1200 mg were down titrated to 800 mg for 1 week and then down-titrated to 400 mg for 1 week and subjects in the placebo group received placebo QD for 2 weeks. During Part I, 1 to 2 concomitant AEDs were allowed in this study and were to be kept stable during the course of the study.

ELIGIBILITY:
Inclusion Criteria

At V1 (screening), patient must be/have:

1. Written informed consent signed by patient.
2. Aged 16 years or more (patients under 18 years of age require parental/legal representative consent). In North America as well as in other participating countries, when appropriate and/or required by state or local law, minor patients must give written informed assent prior to participation in the study.
3. A documented diagnosis of epilepsy since at least 12 months prior to screening.
4. At least 4 partial-onset seizures (including subtypes of simple partial, complex partial and partial seizures evolving to secondarily generalised) on the 4 weeks prior to screening.
5. Currently treated with 1 or 2 AEDs (any except OXC), in a stable dose regimen during at least 1 month prior to screening. Patients using vigabatrin should have been on this medication for at least 1 year with no deficit in visual field identified (a confirmatory test should be available within 1 month before study entry). The device for VNS should be implanted at least 6 months before screening; parameters need to be stable for at least 1 month prior to screening (VNS will not be counted as concomitant AED).
6. Excepting epilepsy, patient is judged to be in general good health based on medical history, physical examination findings, and clinical laboratory test results.
7. Post-menopausal or otherwise incapable of becoming pregnant by reason of surgery or tubal ligation. In case of women of childbearing potential (WOCBP), patient must present a serum beta-human chorionic gonadotropin (B-hCG) test consistent with a non gravid state and agree to remain abstinent or use reliable contraception (hormonal contraception should be combined with a barrier method) beginning at screening and continuing at least to the PSV.

   At V2 (randomisation), patient must have:
8. At least 8 partial-onset seizures during baseline with at least 3 partial-onset seizures in each 4-week section of the 8-week baseline period prior to randomisation (documented in a diary) and no seizure-free interval exceeding 28 consecutive days.
9. In case of WOCBP, patient must present a urine B-hCG test consistent with a non gravid state.
10. Diaries satisfactorily completed by the patient or his/her caregiver.
11. Satisfactorily complied with the study requirements during the baseline period (including no changes in concomitant AED therapy should have occurred in the baseline period).

Exclusion Criteria

At V1 (screening), patients must not be/have:

1. Only simple partial seizures with no motor symptomatology (classified as A2 4 according to the International Classification of Epileptic Seizures).
2. Primarily generalised seizures.
3. Known progressive neurological disorders (progressive brain disease; epilepsy secondary to progressive cerebral lesion).
4. Occurrence of seizures too close to count accurately.
5. History of status epilepticus or cluster seizures (i.e., 3 or more seizures within 30 minutes) within the 3 months prior to screening.
6. Seizures of non-epileptic origin.
7. Seizures of psychogenic origin within the last 2 years.
8. Major psychiatric disorders.
9. Documented diagnosis of schizophrenia with accompanying documented history of at least 1 acute psychosis episode within the last 2 years) or history of suicide attempt.
10. Currently treated with OXC.
11. Using benzodiazepines on more than an occasional basis (defined as more than 2 times per week), except when used chronically as AED.
12. Known exposure to Eslicarbazepine acetate from previous study.

    o Previous use of Eslicarbazepine acetate or participation in a clinical study with Eslicarbazepine acetate (patients not exposed to Eslicarbazepine acetate [e.g., screen failed] are allowed).
13. Known hypersensitivity to carboxamide derivatives.
14. History of abuse of alcohol, drugs or medications within the last 2 years.
15. Uncontrolled cardiac, renal, hepatic, endocrine, gastrointestinal, metabolic, haematological or oncology disorder.
16. Second or third-degree atrioventricular blockade not corrected with a pacemaker.
17. Relevant clinical laboratory abnormalities (e.g., sodium <130 mmol/L, alanine or aspartate transaminases >2.0 times the upper limit of the normal, white blood cell [WBC] count <3,000 cells/mm3) or for patients of Asian ancestry, positive HLA B*1502 test.
18. Estimated creatinine clearance <60 mL/min [men: (140-age) x weight/serum creatinine x 72; women: (0.85) (140-age) x weight/serum creatinine x 72. Age in years, weight in kg, and serum creatinine in mg/dL].
19. Pregnant or nursing.
20. Participation in other drug clinical trial within the last 2 months or received an investigational drug within 5 half-lives of this other product, whichever is longer. Patient(s) who are known to have not taken any doses of study drug(s) in earlier study(ies) (e.g. screen-failures) are allowed without any time limitation.
21. Not ensured capability to perform the trial.
22. Any other condition or circumstance that, in the opinion of the Investigator, may compromise the patient's ability to comply with the study protocol.
23. Currently treated with VNS, but implanted <6 months before screening or parameters not stable for at least 1 month prior to screening.

    At V2 (randomisation), patients must not be/have:
24. Inadequate compliance to concomitant AEDs during the 8-week baseline period or to screening exclusion criteria.
25. Inadequate completion of the study diary.
26. Any other condition or circumstance that, in the opinion of the Investigator, may compromise the patient's ability to comply with the study protocol.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 653 (Actual)
Dates: Start 2008-12-02; Primary Completion 2012-01-12 (Actual); Study Completion 2012-01-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (162):
- United States (106):
  - University of South Alabama Department of Neurology, Mobile, Alabama
  - Neurology Clinic, P.C., Northport, Alabama
  - 21st Century Neurology - Division of Xenoscience, Inc., Phoenix, Arizona
  - Barrow Neurological Institute / St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Phoenix Neurological Associates/Clinical Research Advantage, Phoenix, Arizona
  - ANI Research, PC, Sun City, Arizona
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Neurology, Conway, Arkansas
  - Clinical Trials Inc., Little Rock, Arkansas
  - Kern County Neurological Medical Group, INC., Bakersfield, California
  - Neuro-Pain Medical Center, Inc., Fresno, California
  - Loma Linda University, Loma Linda, California
  - Collaborative Neuroscience Network, INC, Long Beach, California
  - Viking Clinical Research Center, Murrieta, California
  - Bright Minds Institute, San Francisco, California
  - Milestone Clinical Research, San Jose, California
  - Neurosearch II, Inc., Ventura, California
  - University of Colorado Health Sciences, Aurora, Colorado
  - Denver Health, Denver, Colorado
  - Bradenton Research Center, Bradenton, Florida
  - Optima Neurological Services, LLC, Gainesville, Florida
  - University of Florida Department of Neurology, Gainesville, Florida
  - NW FL Clinical Research Group, LLC, Gulf Breeze, Florida
  - Palm Springs Research Institute, Hialeah, Florida
  - University of Florida, Jacksonville, Florida
  - Pharmax Research Clinic, Miami, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - University of Miami - Miller School of Medicine Department of Neurology, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Neuroscience Consultants, Miami, Florida
  - Kendall South Medical Center, Inc., Miami, Florida
  - Medsol Clinical Research Center, Port Charlotte, Florida
  - Lovelace Scientific Resources, Sarasota, Florida
  - University of South Florida - Department of Neurology, Tampa, Florida
  - Pediatric Epilepsy & Neurology Specialists, PA, Tampa, Florida
  - Lovelace Scientific Resources, Venice, Florida
  - Palm Beach Clinical Research Network, LLC., Wellington, Florida
  - Harbin Clinic, Rome, Georgia
  - Consultants in Epilepsy and Neurology, PPLC, Boise, Idaho
  - Southern Ilinois University School of Medicine, Springfield, Illinois
  - Josephson Wallack Munshower Neurology P.C., Indianapolis, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - University of Kentucky, Lexington, Kentucky
  - LSUHSC Epilepsy Center, New Orleans, Louisiana
  - Louisiana Research Associates, Inc., New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Mid-Atlantic Epilepsy and Sleep Centre, Bethesda, Maryland
  - MGH Epilepsy Service Massachusetts, General Hospital, Boston, Massachusetts
  - Wayne State University/Detroit Medical Center, Detroit, Michigan
  - Minneapolis Clinic of Neurology, Ltd, Golden Valley, Minnesota
  - Minnesota Epilepsy Group, P.A., Saint Paul, Minnesota
  - Precise Research Centers, Flowood, Mississippi
  - The Comprehensive Epilepsy Care Centre for Chidren and Adults, Chesterfield, Missouri
  - The Cooper Health System, Camden, New Jersey
  - Clinical Research Centre of New Jersey, Gibbsboro, New Jersey
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - UMDNJ-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - St. Joseph Regional Medical Center, Paterson, New Jersey
  - Shore Neurology, PA, Toms River, New Jersey
  - Albany Medical College - Neurosciences Institute, Albany, New York
  - Five Towns Neuroscience Research, Cedarhurst, New York
  - Neurological Care of CNY, Liverpool, New York
  - Beth Israel Medical Center, New York, New York
  - NYU Comprehensive Epilepsy Centre, New York, New York
  - Wiell Cornell Medical Centre Epilepsy Centre, New York, New York
  - Dent Neurologic Institute, Orchard Park, New York
  - Strong Epilepsy Center - University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - The Neurological Institute, P.A., Charlotte, North Carolina
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - Wilmington Medical Research, Wilmington, North Carolina
  - Ohio State University Medical Centre, Columbus, Ohio
  - Neurology Specialists, Inc, Dayton, Ohio
  - University of Toledo - Health Science Campus, Toledo, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Tulsa Clinical Reserch, Tulsa, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Comprehensive Epilepsy Center - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University School of Medicine - Department of Neurology, Philadelphia, Pennsylvania
  - Childrens Hospital of Pittsburg of UPMC - Division of Child Neurology, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Private Practice of Dr. Edwin Green, Brownwood, Texas
  - Texas Neurology, PA, Dallas, Texas
  - Neurology Consultants of Dallas, P.A., Dallas, Texas
  - Neurological Clinic of Texas, Dallas, Texas
  - UTSWMC Department of Neurology, Division of Epilepsy Research, Dallas, Texas
  - Medistat Clinical Research, DeSoto, Texas
  - Nemmar Clinical Resources, DeSoto, Texas
  - Houston Neurology and Sleep Center, Houston, Texas
  - Innovative Clinical Trials, San Antonio, Texas
  - Road Runner Research, San Antonio, Texas
  - Scott and White Memorial Hospital Sherwood and Brindley Foundation, Temple, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - University of Virginia - Comprehensive Epilepsy Program, Charlottesville, Virginia
  - Sentara Medical Group, Neurology Specialists Sentara Heart Hospital, Norfolk, Virginia
  - Neurological Associates of Washington/Clinical Trials of America, Inc, Bellevue, Washington
  - Ranier Clinical Research Center, Renton, Washington
  - University Washington Regional Epilepsy Center Harborview, Seattle, Washington
  - MultiCare Adult Neurology, Tacoma, Washington
  - Dean & St. Mary's Outpatient Center Neurological Institute and Spine Center, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Regional Epilepsy Centre of Aurora Healthcare- St. Luke's Medical Centre, Milwaukee, Wisconsin
  - Medical College of Wisconsin - Department of Neurology, Milwaukee, Wisconsin
- Argentina (10):
  - Hospital Privado de la comunidad de Mar de Plata, Buenos Aires
  - CEMIC, Buenos Aires
  - Centro Neurológico de Tratamiento y Rehabilitación, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Ramos Mejía, Capital Federal
  - Hospital Británico, Capital Federal
  - Fleni, Capital Federal
  - Instituto Médico Especializado (IME), Capital Federal
  - Hospital Privado - Centro Médico de Córdoba S.A., Córdoba
  - Centro de Neurologia y Neurorehabilitacion, Córdoba
- Belgium (3):
  - Centre Neurologique William Lennox, Ottignies
  - Clinique Saint-Pierre, Ottignies
  - AZ. Sint-Augustinus, Wilrijk
- Brazil (10):
  - Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte
  - Hospital das Clínicas - UNICAMP, Campinas
  - Instituto de Neurologia de Curitiba, Curitiba
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Hospital São Lucas - PUCRS, Porto Alegre
  - Hospital das Clinicas da FMRP, Ribeirão Preto
  - Faculdade de Medicina do ABC, Santo André
  - Irmandade da Santa Casa de Misericórdia de São Paulo, São Paulo
  - Hospital Brigadeiro, São Paulo
  - Hospital São Paulo - UNIFESP, São Paulo
- Canada (3):
  - University of Calgary Clinical Neurosciences, Calgary, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- The Cyprus Institute of Neurology, Nicosia, Cyprus
- France (8):
  - CENTRE HOSPITALIER PELLEGRIN, CHU de BORDEAUX, Bordeaux
  - Hopital Femme-Mere-Enfant, Hospices Civils de Lyon, Bron
  - Hopital Roger Salengro, Chru de Lille, Lille
  - Hopital Gui de Chauliac, Chu de Montpellier, Montpellier
  - Hopital Central, Chu de Nancy, Nancy
  - Centre Hospitalier Sainte-Anne, Paris
  - Hopital Pontchaillou, Chru de Rennes, Rennes
  - Hopital Civil, Chru de Strasbourg, Strasbourg
- Germany (5):
  - Epilepsie-Zentrum Berlin Brandenburg am Evangelischen Krankenhaus Königin Elisabeth Herzberge, Berlin
  - Charite, Universitätsmedizin Berlin, CVK, Berlin
  - Universitätsklinikum Essen, Essen
  - Klinik für Neurologie, Klinische Neurophysiologie und Stroke Unit, Munich
  - Klinik und Poliklinik für Neurologie der Universität Regensburg im Bezirksklinikum, Regensburg
- Greece (3):
  - Evangelismos General Hospital, Athens
  - Agios Loukas (St. Luke's) Hospital, Thessaloniki
  - General Hospital of Thessaloniki "Papanikolaou", Thessaloniki
- Italy (7):
  - Azienda Ospedaliero, Universitaria "Ospedali Riuniti", Clinica della Malattie del Sistema Nervoso, Università di Foggia, Foggia
  - A.O.U Policlinico di Messina, Messina
  - Università degli Studi di Napoli Policlinico Federico II, Napoli
  - Azienda Ospedaliero - Universitaria Maggiore della Carità, Novara
  - Istituto Neurologico Casimiro Mondino, Pavia
  - Università Cattolica del Sacro Cuore Policlinico "A. Gemelli", Roma
  - Azienda Universitatia Ospedaliera San Giovanni Battista, Torino
- Poland (6):
  - Centrum Neurologii Klinicznej, Krakow
  - NZOZ Polimedica, Lodz
  - Wojewódzki Szpital Specjalistyczny w Lublinie Oddzial Neurologii, Lublin
  - Wojewódzki Szpital Specjalistyczny w Olsztynie, Oddzial Neurologii, Olsztyn
  - NZOZ "NEURO - KARD,"Ilkowski I Partnerzy Spólka, Partnerska Lekarzy, Poznan
  - Instytut Psychiatrii i Neurologii, II Klinika Neurologiczna, Warsaw

REFERENCES:
- [Derived] Andermann E, Rosenfeld W, Penovich P, Rogin J, Cendes F, Carreno M, Ramsay RE, Ben-Menachem E, Gama H, Rocha F, Soares-da-Silva P, Tosiello R, Blum D, Grinnell T. Comparative analysis of the safety and tolerability of eslicarbazepine acetate in older (>/=60 years) and younger (18-59 years) adults. Epilepsy Res. 2021 Jan;169:106478. doi: 10.1016/j.eplepsyres.2020.106478. Epub 2020 Oct 10. PMID 33338829
- [Derived] Cramer JA, Colman S, Anastassopoulos KP, Grinnell T, Mehta D, Williams GR. Associations between seizure severity change and patient characteristics, changes in seizure frequency, and health-related quality of life in patients with focal seizures treated with adjunctive eslicarbazepine acetate: Post hoc analyses of clinical trial results. Epilepsy Behav. 2020 Nov;112:107312. doi: 10.1016/j.yebeh.2020.107312. Epub 2020 Aug 12. PMID 32801102

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 173 investigational sites in 19 countries (North America, 89 sites; Rest-of-World [ROW], 84 sites) screened and enrolled subjects. Of these, 160 sites randomized subjects into the study.
  Studied period (years):
  * First subject first visit: 02 December 2008
  * Last subject last visit: 12 January 2012 (Part I)
Pre-assignment Details: The first period was an 8-week observation baseline period (Week -8 to Week -1) during which subjects were instructed on how to complete the seizure diary. At the end of the 8 week observational baseline period, eligible subjects were randomized in a 1:1:1 allocation ratio to 1 of 3 treatment groups (with a blinded treatment assignment)
Groups:
- Placebo: Matching placebo tablets QD orally
- 800 mg QD; 1200 mg QD: The study drug was a conventional immediate-release tablet of eslicarbazepine (ESL) and provided as either 400 mg or 800 mg dosage strengths (the 800 mg tablets were not used in North America). The composition was directly proportional between the strengths. The excipients used were standard pharmaceutical excipients of compendial grade, widely used in the pharmaceutical industry. The medication was taken orally.
Period: Overall Study
Arm/Group | Placebo | 800 mg QD | 1200 mg QD
Started | 226 | 216 | 211
Safety Population | 224 | 216 | 210
Intention-to-treat (ITT) Population | 220 | 215 | 205
Completed | 189 | 173 | 142
Not Completed | 37 | 43 | 69
Not completed — Adverse Event | 9 | 21 | 45
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Non-Compliance with Study Drug | 5 | 1 | 3
Not completed — Physician Decision | 1 | 0 | 3
Not completed — Pregnancy | 2 | 1 | 0
Not completed — Protocol Violation | 4 | 3 | 3
Not completed — Withdrawal by Subject | 7 | 7 | 12
Not completed — Administrative Reasons | 1 | 2 | 1
Not completed — other reasons | 8 | 8 | 1

BASELINE CHARACTERISTICS:
Population: Data Sets Analyzed: Safety Population (all randomized subjects who received at least one dose of study drug after randomization)
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 800 mg QD | 1200 mg QD | Total
Number analyzed (Participants) | 224 | 216 | 210 | 650
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 2 | 6 | 11
  Between 18 and 65 years | 218 | 211 | 202 | 631
  >=65 years | 3 | 3 | 2 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 107 | 105 | 324
  Male | 112 | 109 | 105 | 326
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 46 | 41 | 39 | 126
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 8 | 8 | 24
  White | 142 | 137 | 134 | 413
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 28 | 30 | 29 | 87

OUTCOME MEASURES:

1. Primary Outcome: Seizure Frequency Over the 12-week Maintenance Period.
Time Frame: 12-week maintenance period (Week 3 to week 14)
Population: Intent-to-treat (ITT) population was the primary population for the analysis of efficacy; ITT included all randomized subjects who received at least one dose of study treatment after randomization and had at least one post-baseline seizure frequency assessment.
Measure: Least Squares Mean (Standard Error); unit: Nº Standardized Seizures by 4 weeks
Groups:
- Placebo (ITT Population): Matching placebo tablets QD orally
- ESL 800 mg QD (ITT Population); ESL 1200 mg QD (ITT Population): Oral tablets provided as either 400 mg or 800 mg dosage strengths
Arm/Group | Placebo (ITT Population) | ESL 800 mg QD (ITT Population) | ESL 1200 mg QD (ITT Population)
Number analyzed (Participants) | 220 | 215 | 205
Nº Standardized Seizures by 4 weeks | 7.88 (0.49) [6.98 to 8.90] | 6.54 (0.41) [5.77 to 7.40] | 6.00 (0.40) [5.26 to 6.84]
Statistical Analysis 1: Comparison: Placebo (ITT Population) vs ESL 800 mg QD (ITT Population); Test type: Superiority or Other; p = 0.058, ANCOVA
Statistical Analysis 2: Comparison: Placebo (ITT Population) vs ESL 1200 mg QD (ITT Population); Test type: Superiority or Other; p = 0.004, ANCOVA

2. Secondary Outcome: Proportion of Responders
Description: Subjects who had at least a 50% reduction from baseline in standardized seizure frequency during the maintenance period were classified as responders.
Time Frame: Baseline (Week-8 through Week -1) and Maintenance period (Week 3 to week 14)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | ESL 800 mg QD (ITT Population) | ESL 1200 mg QD (ITT Population)
Number analyzed (Participants) | 220 | 215 | 205
percentage of participants | 23.1 [17.6 to 29.4] | 30.5 [24.2 to 37.4] | 42.6 [35.4 to 50.1]
Statistical Analysis 1: Comparison: Placebo vs ESL 800 mg QD (ITT Population); Test type: Superiority or Other; p = 0.068, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs ESL 1200 mg QD (ITT Population); Test type: Superiority or Other; p = 0.001, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were monitored for the duration of the study, starting at V1
Groups:
- Placebo (Safety Population): Matching placebo tablets QD orally
- ESL 800 mg QD (Safety Population); ESL 1200 mg QD (Safety Population): Oral tablets provided as either 400 mg or 800 mg dosage strengths
Arm/Group | Placebo (Safety Population) | ESL 800 mg QD (Safety Population) | ESL 1200 mg QD (Safety Population)
Serious Adverse Events (participants affected / at risk) | 7/224 | 14/216 | 3/210
Other Adverse Events (participants affected / at risk) | 125/224 | 145/216 | 163/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Safety Population) (N=224) | ESL 800 mg QD (Safety Population) (N=216) | ESL 1200 mg QD (Safety Population) (N=210)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Malaria (Infections and infestations) | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 1
Anticonvulsant drug level below therapeutic (Investigations) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cerebellar syndrome (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 1 | 0
Partial seizures (Nervous system disorders) | 0 | 2 | 0
Partial seizures with secondary generalisation (Nervous system disorders) | 0 | 2 | 0
Simple partial seizures (Nervous system disorders) | 0 | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Safety Population) (N=224) | ESL 800 mg QD (Safety Population) (N=216) | ESL 1200 mg QD (Safety Population) (N=210)
Dizziness (Nervous system disorders) | 19 | 34 | 55
Somnolence (Nervous system disorders) | 12 | 16 | 36
Nausea (Gastrointestinal disorders) | 11 | 16 | 32
Headache (Nervous system disorders) | 17 | 20 | 24
Vomiting (Gastrointestinal disorders) | 3 | 6 | 23
Diplopia (Eye disorders) | 4 | 14 | 22
Vertigo (Ear and labyrinth disorders) | 1 | 6 | 15
Fatigue (General disorders) | 6 | 8 | 11
Sinus bradycardia (Cardiac disorders) | 0 | 4 | 2
Hypothyroidism (Endocrine disorders) | 3 | 4 | 4
Vision blurred (Eye disorders) | 2 | 10 | 9
Visual impairment (Eye disorders) | 1 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1 | 4
Constipation (Gastrointestinal disorders) | 3 | 6 | 4
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 3
Hypoaesthesia oral (Gastrointestinal disorders) | 2 | 1 | 2
Toothache (Gastrointestinal disorders) | 2 | 0 | 4
Asthenia (General disorders) | 3 | 4 | 7
Gait disturbance (General disorders) | 1 | 3 | 3
Irritability (General disorders) | 1 | 4 | 1
Oedema peripheral (General disorders) | 2 | 2 | 2
Pyrexia (General disorders) | 2 | 1 | 4
Influenza (Infections and infestations) | 6 | 4 | 1
Nasopharyngitis (Infections and infestations) | 8 | 6 | 3
Pharyngitis (Infections and infestations) | 3 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 2
Urinary tract infection (Infections and infestations) | 4 | 6 | 4
Contusion (Injury, poisoning and procedural complications) | 4 | 2 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 3 | 1
Head injury (Injury, poisoning and procedural complications) | 2 | 3 | 3
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 2
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 2
Skin laceration (Injury, poisoning and procedural complications) | 2 | 3 | 1
Thermal burn (Injury, poisoning and procedural complications) | 3 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 2
Blood sodium decreased (Investigations) | 0 | 1 | 4
Weight increased (Investigations) | 2 | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 3 | 5 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 4 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 7 | 1
Bone metabolism disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1
Amnesia (Nervous system disorders) | 0 | 3 | 2
Ataxia (Nervous system disorders) | 0 | 4 | 10
Balance disorder (Nervous system disorders) | 1 | 7 | 8
Cerebellar syndrome (Nervous system disorders) | 0 | 1 | 2
Coordination abnormal (Nervous system disorders) | 0 | 1 | 3
Disturbance in attention (Nervous system disorders) | 2 | 0 | 2
Dysarthria (Nervous system disorders) | 0 | 3 | 8
Dyskinesia (Nervous system disorders) | 0 | 0 | 2
Lethargy (Nervous system disorders) | 1 | 0 | 2
Memory impairment (Nervous system disorders) | 1 | 1 | 2
Migraine (Nervous system disorders) | 1 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 6
Nystagmus (Nervous system disorders) | 0 | 0 | 6
Partial seizures (Nervous system disorders) | 7 | 6 | 4
Partial seizures with secondary generalisation (Nervous system disorders) | 1 | 3 | 0
Tremor (Nervous system disorders) | 1 | 4 | 9
Anxiety (Psychiatric disorders) | 5 | 6 | 1
Depression (Psychiatric disorders) | 6 | 5 | 6
Insomnia (Psychiatric disorders) | 2 | 4 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 4
Flushing (Vascular disorders) | 0 | 1 | 2
Hypertension (Vascular disorders) | 5 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other